CLINICAL TRIAL: NCT02102295
Title: Clinical Study of an Ascorbic Acid Derivative Dentifrice in Patients With Gingivitis
Brief Title: Effects of Antioxidant Dentifrice on Gingivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lion Corporation (Industry)
Collaborators: Osaka University (Other); Tohoku University (Other); Nihon University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LionSDP-6
Record Dates: First submitted 2014-03-23; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Gingivitis
Keywords: Gingivitis; antioxidant; dentifrice; Ascorbic Acid Derivative; L ascorbic acid 2 phosphate magnesium salt
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental toothpaste (Active Comparator): L-ascorbic acid 2-phosphate magnesium salt / fluoride
  Interventions: Drug: Experimental toothpaste
- Control toothpaste (Placebo Comparator): fluoride
  Interventions: Drug: Control toothpaste

INTERVENTIONS:
Drug: Experimental toothpaste — Experimental toothpaste was containing 0.3% L-ascorbic acid 2-phosphate magnesium salt and 950 ppm fluoride. The registered participants were instructed to brush their teeth twice a day in their customary manner.
  Other Names: L-ascorbic acid 2-phosphate magnesium salt toothpaste
  Arms: Experimental toothpaste
Drug: Control toothpaste — Control toothpaste was containing 950 ppm fluoride. The registered participants were instructed to brush their teeth twice a day in their customary manner.
  Other Names: Fluoride toothpaste
  Arms: Control toothpaste

SUMMARY:
The purpose of this study is to investigate the effect of a dentifrice containing L-ascorbic acid 2-phosphate magnesium salt on gingival inflammation, gingival bleeding and gingival redness.

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥ 20 and < 65 y with at least 16 permanent teeth.
* Gingival inflammation or mean baseline GI ≥ 0.5 without severe periodontal disease enough to require professional therapy.
* Written informed consent to participate.

Exclusion Criteria:

* Taking medications that could influence periodontal tissue health, such as antimicrobials and antihypertensives within 1 month before starting the trial.
* Use of orthodontic appliances.
* Pregnancy or planning to become pregnant during the trial period.
* Previous participation in any other clinical trial.
* Inability of patient to understand the study purpose and/or study protocols.
* Judged unsuitable by investigators for other reasons.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Gingival Index | 3 months

SECONDARY OUTCOMES:
Gingivitis Severity Inedex | 3 months
Gingival Redness | 3 months
  Gingival redness was measured as an indicator of the degree of local chromatic changes in the gingiva.

OTHER OUTCOMES:
salivary antioxidant status | 3 months
  Salivary antioxidant status was assessed by the ferric reduction ability of plasma (FRAP).

CONTACTS AND LOCATIONS:
Overall Officials: Shinya Murakami, Principal Investigator — Osaka University
Locations (4):
- Japan (4):
  - Nihon University Hospital, School of Dentistry at Matsudo, Matsudo, Chiba
  - Tohoku University Dental Hospital, Sendai, Miyagi
  - Osaka University Dental Hospital, Suita, Osaka
  - Nihon University Dental Hospital, Chiyoda-ku, Tokyo

REFERENCES:
- [Derived] Shimabukuro Y, Nakayama Y, Ogata Y, Tamazawa K, Shimauchi H, Nishida T, Ito K, Chikazawa T, Kataoka S, Murakami S. Effects of an ascorbic acid-derivative dentifrice in patients with gingivitis: a double-masked, randomized, controlled clinical trial. J Periodontol. 2015 Jan;86(1):27-35. doi: 10.1902/jop.2014.140138. PMID 25277459